CLINICAL TRIAL: NCT00382954
Title: A Phase I Study Using Bortezomib (Velcade, Formerly Known as PS-341) With Weekly Idarubicin for the Treatment of Elderly (>/= 60 Years) and Relapsed Patients With Acute Myelogenous Leukemia
Brief Title: Phase I Using Velcade & Idarubicin in Elderly and Relapsed AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Dianna Howard, MD, University of Kentucky
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-BMT-145
Record Dates: First submitted 2006-09-28; First posted 2006-10-02 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Acute Myelogenous Leukemia; AML; Relapse; Elderly; Velcade; Idarubicin; Bortezomib
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Bortezomib; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase 1 escalation (Experimental)
  Interventions: Drug: Velcade; Drug: Idarubicin

INTERVENTIONS:
Drug: Velcade — velcade (4 original dosing levels with 3 modified dosing levels) I.V. on days 1, 4, 8, 11, 15, 18, 22, and 25 for 4 weeks concurrent with the Idarubicin
  Other Names: Bortezomib
Drug: Idarubicin — I.V., 8, or 10 or 12 mg/m^2 weekly (days 1, 8, 15, and 22) for 4 weeks

SUMMARY:
The purpose of this study is to determine the maximal tolerated dose (MTD) of bortezomib and idarubicin given in combination to newly diagnosed AML patients >60 years or relapsed AML patients.

Another purpose of this study is to determine the dose limiting toxicities associated with bortezomib in combination with idarubicin in newly diagnosed AML patients >60 years or relapsed AML patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: > 60 years of age for newly diagnosed/transformed disease; > 18 years of age for relapsed disease.
* AML with or without antecedent hematologic disorder diagnosed by morphologic, histochemical, or cell surface marker criteria - as defined by the WHO classification (17).
* Newly diagnosed, elderly patients who are considered unsuitable for intensive chemotherapy induction -- antecedent hematologic disorders, pre-existing myelodysplasia, trilineage dyspoiesis, unfavorable cytogenetics, or pre-existing comorbidities.
* Untreated conditions meeting criteria the first and third criteria or patients with diagnosis as in criteria 2 who have relapsed after at least one successful induction therapy. (Relapsed patients treated on this protocol will be patients without a suitable donor for transplant or for whom transplant is not an option for other reasons.)
* Karnofsky performance status >60.
* Adequate cardiac function as evidenced by an ejection fraction on MUGA >/= 40, as well as no evidence of uncontrolled hypertension, New York Heart Class III/IV congestive heart failure, angina pectoris, or ventricular dysrhythmias.
* Adequate renal function as evidenced by a calculated creatinine clearance >/= 30ml/min (Cockcroft-Gault formula).
* Adequate pulmonary function as evidenced by room air and exercise saturations >/= 92 or DLCO >/= 40% or FEV1 >/= 60% of predicted.
* Adequate liver function as evidenced by SGOT/SGPT less than 5 times the ULN and total Bilirubin less than 2 times the ULN except where abnormalities are directly attributable to leukemia.
* Adequate neurologic function -- patients must be currently free of active CNS leukemia as evidenced by cytospin of CSF from lumbar puncture if there is any clinical suspicion for CNS leukemia. As well, patients must not have >/= grade 2 neuropathy by NCI common toxicity criteria (CTC), Version 3.0.
* Prior anthracycline dose in relapsed patients must not exceed 72 mg/m^2 of idarubicin or any dose equivalent to 300 mg/m^2 of adriamycin.
* Patients must be informed and sign a written consent.

Exclusion Criteria:

* Patients with acute promyelocytic leukemia. Patients with uncontrolled systemic infection.
* Patients who are known to be HIV seropositive.
* Patients with evidence of CNS leukemia.
* Patients who are pregnant or lactating.
* Patients with primarily refractory disease unresponsive to a standard induction regimen.
* Patients with a new diagnosis as per inclusion criteria 2, but for whom standard induction chemotherapy would be expected to be well tolerated and a preferred option in the opinion of the principal investigator.
* Patients with relapsed AML, but for whom a suitable donor of stem cells exists and in whom high-dose chemotherapy with hematopoietic stem cell transplant is felt to be a better immediate alternative.
* Patients with any clinically significant abnormality in screening blood chemistry, hematology or urinalysis results that, in the judgment of the investigator, would impede adequate evaluation of adverse events and/or response to treatment, or that requires aggressive intervention.
* Patients with hypersensitivity to Bortezomib, boron, or mannitol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2004-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of bortezomib & idarubicin given in combination, with idarubicin given once weekly for 4 consecutive weeks & bortezomib given twice weekly over the same time. | week 4
Dose limiting toxicities associated with bortezomib in combination with idarubicin. | week 4

SECONDARY OUTCOMES:
Response to the combination of Idarubicin and Bortezomib. | Days 18 & 50
Pre- & post-treatment inhibition of NF-kB activity in the malignant & normal hematopoietic cell populations. | 24 hours after the initial dose of Bortezomib
Induction of p53 levels in the malignant cell populations. | 2 and 24 hours post day +1 Bortezomib
Bortezomib PK when administered to patients with acute leukemia receiving concomitant medications that could lead to drug interactions. In the case of altered pharmacokinetics, a pharmacodynamic assay to check proteasome inhibition may also be applied. | Days 1, 4, 8, 11, 15
Idarubicin PK in order to observe any alteration in metabolism/elimination of Idarubicin & its active metabolite idarubicinol when it is combined with Bortezomib. | Days 1, 4, 8, 11, 15

CONTACTS AND LOCATIONS:
Overall Officials: Dianna Howard, MD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - University of Rochester, Rochester, New York

REFERENCES:
- [Derived] Howard DS, Liesveld J, Phillips GL 2nd, Hayslip J, Weiss H, Jordan CT, Guzman ML. A phase I study using bortezomib with weekly idarubicin for treatment of elderly patients with acute myeloid leukemia. Leuk Res. 2013 Nov;37(11):1502-8. doi: 10.1016/j.leukres.2013.09.003. Epub 2013 Sep 8. PMID 24075534
- See also: University of Kentucky Markey Cancer Center Clinical Trials Listing — http://markey.uky.edu/studysearch